CLINICAL TRIAL: NCT01264666
Title: Phase I Study of Chinese Tea Flavor Liquor on Human Health
Brief Title: Postprandial Effect of Chinese Tea Flavor Liquor on Selected CVD Risk Factors
Acronym: TFL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Guizhou Meijiao Co., Ltd, China (Unknown)
Responsible Party: Jusheng Zheng, Department of food science of nutrition, Zhejiang University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Acute Chinese liquor study
Record Dates: First submitted 2010-12-21; First posted 2010-12-22 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-05

CONDITIONS: Alcohols; Cardiovascular Diseases
Keywords: Chinese tea flavor liquor; postprandial; uric acid; high-sensitive C-reactive protein
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chinese tea flavor liquor (Experimental)
  Interventions: Dietary Supplement: Chinese tea flavor liquor
- Water (Placebo Comparator): Water combined with meal as control.
  Interventions: Dietary Supplement: Water control
- Chinese Meijiao Liquor (Placebo Comparator)
  Interventions: Dietary Supplement: Chinese Meijiao liquor

INTERVENTIONS:
Dietary Supplement: Chinese tea flavor liquor — 60 mL of Chinese tea flavor liquor (45% alcohol content) is consumed with high-fat meal.
  Arms: Chinese tea flavor liquor
Dietary Supplement: Chinese Meijiao liquor
  Arms: Chinese Meijiao Liquor
Dietary Supplement: Water control
  Arms: Water

SUMMARY:
Background: human studies of Chinese liquor are sparse. we hypothesis that Chinese Tea Flavor liquor may be beneficial to CVD risk factors postprandially.

Design: three-way crossover design with one week wash time.16 young men were included to consume 60mL Chinese tea flavor liquor(45% alcohol content), Chinese Meijiao liquor 45% alcohol content) or water control.Blood samples were collected fasted, 0.5,1,2,4 hours postprandially.

Tested serum indices: lipids, glucose, insulin, hs-CRP, uric acid, liver function parameters.

ELIGIBILITY:
Inclusion Criteria:

* no CVD history or liver disease, healthy young men

Exclusion Criteria:

* smokers

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
serum sample | 4 hours
  blood samples were collected at 0,0.5,1,2,4 hours postprandially to get serum sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food Science of Nutrition, Zhejiang University, Hangzhou, Zhejiang, China